CLINICAL TRIAL: NCT03104257
Title: The Neural Correlates of Cannabis Use
Acronym: Multimodal
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mohini Ranganathan, Associate Professor, Yale University
Other Study IDs: 1308012514; 1R01DA040698-01A1 (NIH)
Record Dates: First submitted 2016-12-22; First posted 2017-04-07 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Cannabis Dependence; Healthy
Keywords: Healthy Control, Cannabis, Dependence
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — When specimens and information are stored, researchers are careful to try to protect your identity from discovery by others. Samples and information will receive a unique code. Other researchers will only receive coded samples and information, and will not be able to link the code to subjects. Strict security safeguards are in place to reduce the chance of misuse or unplanned release of information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (2):
- Cannabis Dependent Subjects: Subjects who are frequent cannabis users
  Interventions: Drug: [11-C]OMAR
- Healthy Controls: Subjects with no current cannabis use
  Interventions: Drug: [11-C]OMAR

INTERVENTIONS:
Drug: [11-C]OMAR — The radiotracer, [11-C]OMAR will be administered at no more than 10 micrograms at the beginning of each PET scan.

SUMMARY:
The purpose of this research study is to determine the temporal course of recovery of CB1R availability and neural oscillations, in cannabis-dependent individuals at baseline, following 48 hour confirmed inpatient abstinence and after four weeks confirmed abstinence. This research will also examine associations between CB1R availability, neural oscillations and cognitive function.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the temporal course of recovery of CB1R availability and neural oscillations, in cannabis-dependent individuals at baseline, following 48 hour confirmed inpatient abstinence and after four weeks confirmed outpatient abstinence (confirmed by tracking creatinine adjusted urine THC-COOH levels). This research will also examine associations between CB1R availability, neural oscillations and cognitive function using [11-C]OMAR PET imaging and electroencephalography.

ELIGIBILITY:
Inclusion Criteria: Cannabis Dependent Subjects

* Current cannabis consumption
* Willing to abstain from cannabis use for four weeks

Inclusion Criteria for Healthy Controls

* No current cannabis consumption

Exclusion Criteria:

* MRI metal exclusions and claustrophobia
* Education completed is less than 12 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Research subjects can be both cannabis-using or non-cannabis using males and females between the ages of 18-65.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2016-12; Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
CB1R availability using [11-C]OMAR PET imaging | Change in CB1R availability from baseline to 48 hours and 28 days
  Change in CB1R availability (e.g. volume distribution).

SECONDARY OUTCOMES:
Changes in Cognition during withdrawal using a computerized battery | Change in CB1R availability from baseline to 48 hours and 28 days
  Changes in cognitive functions such as attention, memory, motor functioning, and processing speed.
Changes in brain rhythms measured by Electroencephalography | Change in CB1R availability from baseline to 48 hours and 28 days
  Changes in electroencephalographic (EEG) brain rhythms related to information processing.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University
Locations (1):
- Conneticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No